CLINICAL TRIAL: NCT07119827
Title: Neuropsychology and Personality: Personality Traits as a Variable in the Recovery of Patients With Acquired Brain Injury
Brief Title: Personality Traits as a Variable in the Recovery of Patients With Acquired Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Universita di Verona (Other)
Collaborators: CRT Montevarchi (Arezzo), Dr. Benedetta Basagni (Unknown); Azienda USL Toscana Sud Est (Other Government); Centro Cardinal Ferrari, Fontanellato, Parma (Unknown); Montecatone Rehabilitation Institute S.p.A., Imola (Italy) (Unknown); Fondazione IRCCS Santa Lucia, Roma, Italy (Unknown); IRCCS Fondazione Don Carlo Gnocchi, Milano (Unknown); Azienda Unita Sanitaria Locale di Piacenza, Italy (Unknown); Azienda Sanitaria dell'Alto Adige (Other); Azienda Ospedaliero, Universitaria Pisana (Other); Azienda Sanitaria Locale CN1 Cuneo (Other Government); Istituto S.Anna Crotone (Unknown); Dr. Navarro Solano Jorghe, MD of the Fondazione Don Carlo Gnocchi Onlus Santa Maria Nascente center (Unknown); Dr. Pasqualone Eugenia MD Fondazione Don Carlo Gnocchi Onlus of La Spezia center (Unknown); SO Riabilitazione Neuromotoria, IRCCS Fondazione Don Carlo Gnocchi (Firenze) - Francesca Cecchi (Unknown); SO Riabilitazione GCA, IRCCS Fondazione Don Carlo Gnocchi (Firenze) - Bahia Hakiki (Unknown)
Responsible Party: Principal Investigator, Valentina Varalta, Doctor, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 481CET
Record Dates: First submitted 2025-08-05; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ictus; Severe Acquired Brain Injury; sABI
Keywords: premorbid personality; stroke; severe acquired brain injury; recovery; cognitive deficits; motor deficits; disability; psychological functioning; behaviour; sABI
MeSH Terms: conditions — Brain Injuries; Stroke; Cognition Disorders; Neurologic Manifestations; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ischemic or hemorrhagic stroke: Aged between 18 and 80 years; ischemic or hemorrhagic stroke without features of severe acquired brain injury (Glasgow Coma Scale ≥ 8 and no alteration in consciousness); time from onset between 3 and 30 days
  Interventions: Diagnostic Test: Motor, cognitive and psychological assessment
- Severe Acquired Brain Injury (sABI) of traumatic or non-traumatic etiology: Aged between 18 and 80 years; severe Acquired Brain Injury (sABI) of traumatic or non-traumatic etiology meaning that the patient initially presents with a state of coma (Glasgow Coma Scale score < 8) accompanied by simultaneous motor, sensory, cognitive and/or behavioral impairment; Glasgow Coma Scale ≥ 8 and no alteration in consciousness; time from onset between 7 and 90 days; Level of Cognitive Functioning (LCF) >=6
  Interventions: Diagnostic Test: Motor, cognitive and psychological assessment

INTERVENTIONS:
Diagnostic Test: Motor, cognitive and psychological assessment — Participants evaluated at T0 (Initial assessment upon admission to the rehabilitation facility), T1 (at discharge from the inpatient rehabilitation program, as long as at least 30 days have passed since the initial assessment (T0), T2 (at 12 months from the event for patients with stroke, and at 18 months from the event for patients with sABI).

SUMMARY:
This study aims to evaluate the potential effects of premorbid personality on the short- and long-term global cognitive recovery in patients with severe acquired brain injury (sABI) or stroke.

The secondary aims are to assess the effects of premorbid personality on the sort- and long-term recovery in autonomy (disability), cognitive functions, psycho-behavioral functioning, motor skills, and social participation. Evaluate the incidence of premorbid personality alterations. Investigate personality changes 12-18 months after the neurological event.

DETAILED DESCRIPTION:
Participants included in the study will undergo cognitive, motor, psychological, behavioral, personality, and disability assessments at different time points following the neurological event:

T0: Initial assessment upon admission to the rehabilitation facility; within 90 days of the event for patients with severe acquired brain injury (sABI), as soon as cognitive evaluation becomes feasible (LCF ≥ 6); within 30 days of the event for stroke patients, as soon as cognitive assessment is possible.

T1: At discharge from the inpatient rehabilitation program, provided that at least 30 days have passed since the initial assessment (T0).

T2: At 12 months post-event for stroke patients and at 18 months post-event for patients with ABI.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of one of the following two conditions:
* Severe Acquired Brain Injury (sABI) of traumatic or non-traumatic etiology; the term sABI includes acute brain injuries of traumatic or non-traumatic origin (vascular, infectious, metabolic, or anoxic), in which the patient initially presents with a coma state (Glasgow Coma Scale - GCS less than 8) and simultaneously exhibits motor, sensory, cognitive, and/or behavioral impairments.
* Ischemic or hemorrhagic stroke without features of Severe Acquired Brain Injury (sABI) (Glasgow Coma Scale [GCS] score ≥ 8 and no alteration of consciousness).
* Time from injury between:
* 7 and 90 days for Severe Acquired Brain Injury (sABI) patients
* 3 and 30 days for stroke patients
* Level of Cognitive Functioning (LCF) score ≥ 6 for sABI patients
* Signed informed consent for study participation
* Presence of a support family member (caregiver) able to assist with completing the personality questionnaire (HEXACO Adjective Scale, HAS)

Exclusion Criteria:

* Pre-existing neurological pathology
* Severe aphasia or severe inattention that precludes administration of the tests required by the protocol, as identified during cognitive screening.
* Patients with a language barrier due to insufficient proficiency in Italian.
* Particularly vulnerable populations:

The following patients will be excluded from the study: patients in emergency situations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to the Neurorehabilitation Unit (UOC) of AOUI Verona (and collaborating centers) will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | The test is administered (both stroke and sABI) at baseline-T0 (between 3-30 days from onset - ictus; 7-90 days from onset - sABI), at discharge (at least 30 days from T0) and at followup-T2 (12 moths from onset - ictus; 18 months from onset - sABI).
  MoCA is a brief, standardized screening tool designed to detect the global cognitive status of patients. It assesses multiple cognitive domains, including: Attention and concentration, Executive functions, Memory, Language, Visuoconstructional skills, Conceptual thinking, Calculations, Orientation. The test takes approximately 10 to 15 minutes to administer and yields a total score out of 30 points. Higher scores indicates a better performance. In the study it is used to evaluate the potential effects of premorbid personality on the degree of global cognitive rocovery in the short and long term.

SECONDARY OUTCOMES:
Oxford Cognitive Screen (OCS) | The test is administered (both stroke and sABI) at baseline-T0 (between 3-30 days from onset - ictus; 7-90 days from onset - sABI), at discharge (at least 30 days from T0) and at followup-T2 (12 moths from onset - ictus; 18 months from onset - sABI).
  Neuropsychological assessment tool that measures a person's global cognitive status, providing an analysis of key cognitive functions such as memory, executive functions, praxis, attention, language, and visuospatial exploration. Composed of various sub-tests, the OCS allows for the rapid and systematic identification of potential cognitive deficits and is particularly useful in patients with brain damage, such as those with stroke. Higher scores meaning a better performance.
Trial Making Test (TMT) | The test is administered (both stroke and sABI) at baseline -T0 (between 3-30 days from onset - ictus; 7-90 days from onset - sABI), at discharge (at least 30 days from T0) and at followup-T2 (12 moths from onset - ictus; 18 months from onset - sABI).
  Consists of two parts: TMT-A, used as a measure of psychomotor speed and visual search/attention skills; TMT-B used as a measure of attentional set-shifting and mental flexibility. Time needed to complete the tasks is recorded.
Digit Span Forward | The test is administered (both stroke and sABI at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  Digit Span Forward is a brief, standardized subtest used to assess attention and short-term verbal memory. It requires the patient to repeat a sequence of numbers in the same order as presented by the examiner, with increasing length. The task evaluates auditory attention, immediate recall, and working memory span. Higher scores indicate better performance. In the study, it is used to investigate the relationship between premorbid personality traits and specific cognitive functions, particularly attentional capacity.
Corsi Span Forward | The test is administered (both stroke and sABI)at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  Corsi Span Forward is a brief, standardized visuospatial memory task used to assess short-term visuospatial memory and attention. During the task, the examiner taps a sequence of blocks on a board, and the patient is required to reproduce the same sequence in the same order. The length of the sequence increases progressively. Higher scores indicate better visuospatial short-term memory performance. In the study, it is used to explore the association between premorbid personality traits and the recovery of visuospatial attention and memory functions.
Digit Span Backward | The test is administered both stroke and sABI, at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  Digit Span Backward is a standardized neuropsychological task that assesses working memory and attention. In this task, the examiner reads aloud a sequence of digits, and the patient is required to repeat them in reverse order. The sequence length increases progressively until the patient can no longer recall the digits correctly. Higher scores reflect better working memory performance. In the study, it is used to investigate the relationship between premorbid personality traits and recovery of working memory and attentional control.
Corsi span backward | The test is administered both stroke and sABI, at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  Corsi Span Backward is a standardized visuospatial memory task used to assess working memory and executive functions. In this task, the examiner taps a sequence of blocks on a board, and the patient is required to reproduce the sequence in reverse order. The sequences increase in length until the patient can no longer reproduce them correctly. Higher scores indicate better visuospatial working memory and manipulation abilities. In the study, it is used to examine how premorbid personality traits may influence the recovery of executive and visuospatial memory functions.
Rey Auditory Verbal Learning Test (RAVLT) | The test is administered both stroke and sABI, at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  The Rey Auditory Verbal Learning Test (RAVLT) is a standardized neuropsychological assessment of verbal learning and memory. The test involves the oral presentation of a list of 15 unrelated words over five learning trials, followed by immediate recall after each trial, an interference list, immediate recall of the original list, and delayed recall after a 20-30-minute interval. A recognition trial is also included. RAVLT. Higher scores indicate better verbal learning and memory abilities. In the study, it is used to assess how premorbid personality may influence short- and long-term verbal memory recovery.
Test della Figura di Rey - Test della Figura di Taylor | The test is administered both stroke and sABI, at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  The Rey-Osterrieth Complex Figure Test (ROCFT) and the Taylor Complex Figure Test (TCFT) are standardized neuropsychological tools used to assess visuospatial constructional abilities and non-verbal memory. Participants are asked to copy a complex figure (Rey or Taylor) and then reproduce it from memory after a short delay and again after a longer delay. The TCFT is used as an alternative version to minimize learning effects during repeated assessments. These tests evaluate multiple cognitive processes, including visuoperception, planning, attention, working memory, and long-term visuospatial memory. Higher scores reflect better performance. In the study, they are used to evaluate the influence of premorbid personality traits on visuospatial memory and planning skills in the short and long term.
Stroop Test (ST) | The test is administered both stroke and sABI, at baseline-T0 (between 3-30 days from onset - ictus; 7-90 days from onset - sABI), at discharge (at least 30 days from T0) and at followup-T2 (12 moths from onset - ictus; 18 months from onset - sABI).
  Evaluates attention and the ability to inhibit automatic responses. The Stroop effect is evaluated by computing a time interference effect (based on execution time) and an error interference effect (based on number of errors).
Modified Five Point Test (MFPT) | The test is administered (both stroke and sABI) at baseline-T0 (between 3-30 days from onset - ictus; 7-90 days from onset - sABI), at discharge (at least 30 days from T0) and at followup-T2 (12 moths from onset - ictus; 18 months from onset - sABI).
  It measures figural fluency by assessing the ability to initiate mental productivity and self-monitoring during a visual-spatial task. Performance is assessed by scoring the total number of correct and unique designs generated in 3 min (UDs), and the total number of UDs produced into strategies (CSs).
Phonemic fluency | The test is administered (only sABI) at baseline-T0 (between 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 ( 18 months from onset - sABI).
  Phonemic Fluency is a brief verbal task assessing executive functions, especially lexical retrieval and cognitive flexibility. Participants must say as many words as possible beginning with a given letter in 60 seconds. Higher scores reflect better executive functioning. In the study, it assesses the potential impact of premorbid personality on verbal recovery.
Semantic fluency | The test is administered (only sABI) at baseline-T0 (between 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 ( 18 months from onset - sABI).
  Semantic Fluency assesses verbal memory and executive functioning. Participants list as many words as possible from a semantic category (e.g., animals) in 60 seconds. Higher scores indicate better cognitive performance. In the study, it evaluates the influence of premorbid personality on language and executive recovery.
Verbal Reasoning Test (VRT) | Administered at baseline-T0 (3-30 days post-stroke; 7-90 days post-sABI), at discharge (≥30 days from T0), and at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  The Verbal Reasoning Test evaluates verbal reasoning skills through tasks such as identifying absurdities, intruders, relationships, differences, idiomatic expressions, familiarity, and classifications. Higher scores indicate stronger verbal reasoning. In the study, it assesses how premorbid personality influences verbal reasoning recovery.
Brain Injury Rehabilitation Trust questionnaire (BIRT) | Administered (both sABI and stroke) at at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Both versions (for patient, for relatives). Self-report tools used to assess psycho-behavioral functioning in individuals with brain injury. It evaluates emotional, behavioral, and social aspects relevant to rehabilitation outcomes. Higher scores indicate greater difficulties. In the study, it is used to explore the impact of premorbid personality on psycho-behavioral recovery.
Hospital Anxiety and Depression Scale (HADS) | Administered (both stroke and sABI) at baseline-T0 (3-30 days post-stroke; 7-90 days post-sABI), at discharge (≥30 days from T0), and at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Is a self-administered questionnaire designed to assess anxiety and depression symptoms in medically ill patients. It consists of 14 items divided equally between anxiety and depression subscales. Higher scores indicate greater symptom severity. In the study, it is used to evaluate the influence of premorbid personality on psychological well-being during recovery.
HEXACO Adjective Scale (HAS) | Administered (both stroke an sABI) at baseline-T0 (3-30 days post-stroke; 7-90 days post-sABI) and at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Is a self-report personality questionnaire assessing six major personality dimensions: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness, and Openness to Experience. It uses adjective-based items to capture trait levels. Higher scores reflect stronger expression of each trait. In the study, it is used to investigate the role of premorbid personality in cognitive and functional recovery.
Disability Rating Scale (DRS) | Administered at baseline-T0 (3-30 days post-stroke; 7-90 days post-sABI), at discharge (≥30 days from T0), and at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Is a standardized tool used to assess the level of disability and functional changes in individuals with brain injury. It evaluates areas such as consciousness, cognitive ability for self-care, dependence on others, and employability. Scores range from no disability to extreme vegetative state, with higher scores indicating greater disability. In the study, it is used to measure functional recovery and independence over time.
Frenchay Activities Index (FAI) | Administered (both stroke and sABI) at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Is a questionnaire designed to assess the level of participation in instrumental activities of daily living (IADLs) following brain injury or stroke. It evaluates domestic chores, leisure, social activities, and work-related tasks. Higher scores indicate greater independence and activity participation. In the study, it is used to monitor social participation and functional recovery.
Fugl Mayer (FM) | The test is administered both stroke and sABI, at baseline-T0 (between 3-30 days from onset - stroke; 7-90 days from onset - sABI), at discharge (at least 30 days from T0), and at follow-up T2 (12 months from onset - stroke; 18 months from onset - sABI).
  Is a standardized scale used to evaluate motor functioning, balance, sensation, and joint functioning in post-stroke patients. It is widely used to assess recovery of motor impairment, particularly in the upper and lower extremities. Higher scores indicate better motor function. In the study, it is used to measure motor recovery over time.
Motricity Index (MI) | Administered (both stroke and sABI) at baseline-T0 (3-30 days post-stroke; 7-90 days post-sABI), at discharge (≥30 days from T0), and at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Is a clinical scale used to assess motor strength in patients with neurological impairments, especially after stroke. It evaluates muscle power in the upper and lower limbs through specific movements. Higher scores indicate greater muscle strength and motor function. In the study, it is used to monitor motor recovery and functional status.
Modified Ashworth Scale (MAS) | Administered (both stroke and sABI) at baseline-T0 (3-30 days post-stroke; 7-90 days post-sABI), at discharge (≥30 days from T0), and at follow-up T2 (12 months post-stroke; 18 months post-sABI).
  Is a clinical tool used to measure muscle spasticity in patients with neurological conditions such as stroke or brain injury. It assesses resistance during passive soft-tissue stretching and grades spasticity on a scale from 0 (no increase in muscle tone) to 4 (affected part rigid). Higher scores indicate greater spasticity. In the study, it is used to evaluate changes in muscle tone during motor recovery.
Modified barthel Index (MBI) | Administered (only stroke) at baseline-T0 (3-30 days post-stroke), at discharge (≥30 days from T0), and at follow-up T2 (12 months post-stroke; ).
  Is a clinical scale used to measure a patient's level of independence in performing basic activities of daily living (ADLs), such as feeding, bathing, grooming, dressing, bowel and bladder control, mobility, and stair climbing. Higher scores indicating greater functional independence. In the study, it is used to assess disability levels and functional outcomes during rehabilitation.
Disability Rating Scale (DRS) | Administered (only sABI) at baseline-T0 (7-90 days post-sABI), at discharge (≥30 days from T0), and at follow-up T2 (18 months post-sABI).
  Is a clinical tool used to assess the overall level of disability in individuals recovering from severe brain injury, including traumatic and non-traumatic causes. It evaluates a range of functional areas, including consciousness, cognitive ability for self-care, level of dependence, and psychosocial adaptability. Scores range from 0 (no disability) to 29 (extreme vegetative state), with higher scores indicating greater disability. In the study, it is used to monitor functional recovery and global disability over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Sezione medicina fisica e riabilitativa dipartimento di neuroscienze, verona, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: Undecided